CLINICAL TRIAL: NCT02139475
Title: Factors Influencing Quality of Bowel Cleansing for Colonoscopy in Patients With Colorectal Cancer Surgery; Prospective Observational Study
Status: Terminated | Type: Observational
Why Stopped: All the patients who had been targeted were registered.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2013-0772
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2017-12

CONDITIONS: Colorectal Cancer
Keywords: bowel cleansing, colorectal cancer surgery
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Colonoscopy: patients undergoing colonoscopy after colorectal cancer surgery
  Interventions: Procedure: Colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy

SUMMARY:
The aim of this study is to clarify the factors influencing quality of bowel cleansing for colonoscopy in patients with colorectal cancer surgery and confirm the adequate bowel cleaning method for patients with colorectal cancer surgery. Through this, ultimately in patients with a history of colorectal cancer who have high risk of colorectal cancer, it could be possible to detect cancerous lesions early and increase the survival rate.

This study is based on observational study Subjects are the patients with colorectal cancer surgery who visits the out patients clinic for follow-up colonoscopy The patient's medical records on the basis of information collected at the point of the colonoscopy performed Quality of bowel cleansing is calculated with the Boston bowel preparation scale Patient compliance and satisfaction are measured.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 20
* patients who underwent colorectal cancer surgery
* patients who underwent follow-up colonoscopy as a conventional medical procedures

Exclusion Criteria:

* age < 20
* patients who have ileus or bowel obstruction
* patients in pregnant status
* Patients who did not consent to research

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing colonoscopy after colorectal cancer surgery
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2013-12; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Boston bowel preparation scale (BBPS) | 1 hour
  In this scale, the colon is divided in three segments: the right side (including cecum and ascending colon), the transverse colon (including the flexures) and the left sided colon, which includes the descending colon, sigmoid and rectum. Mucosal view should be scored after cleansing maneuvers like suctioning or washing have been performed. For all three sections cleansing is assessed and given a score ranging from 0 to 3. Therefore, the maximum BBPS score for a perfectly clean colon without any residual liquid is 9 and the minimum BBPS score for an unprepared colon is 0. BBPS score ≥6 in considered an adequate bowel preparation.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea